CLINICAL TRIAL: NCT00781573
Title: Study of Optimal Clopidogrel Duration in Patients Receiving Drug Eluting Stents (SCORE Trial)
Acronym: SCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhash Banerjee, Acting chief of Cardiology, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dallas VA IRB #08-048
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Myocardial Infarction
Keywords: Drug Eluting Stent; Clopidogrel; Optimal duration of clopidogrel post DES stent implantation
MeSH Terms: conditions — Myocardial Infarction | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Clopidogrel (75 mg/day) is continued for another year at the completion of the initial year of clopidogrel and aspirin administration post DES implantation
  Interventions: Drug: Clopidogrel
- 2 (No Intervention): Clopidogrel (75 mg/day) is stopped at the completion of the initial year of clopidogrel and aspirin administration post DES implantation

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel, 75 mg QD, for one year
  Arms: 1

SUMMARY:
Although the optimal duration of clopidogrel (an anti-platelet agent) therapy has been established after bare metal stent implantation in the blood vessels of the heart, there is lack of consensus regarding the optimal duration of therapy after implantation of a drug eluting stents (DES). Current American College of Cardiology guidelines recommend clopidogrel use for at least one year in the absence of contraindications after DES implantation, while recognizing that the optimal duration remains unknown. While an extended clopidogrel therapy (that is beyond the current 1 year recommendation) may increase bleeding complication, it may reduce the rates of adverse cardiovascular events like heart attacks and repeat revascularization procedures. A clinical trial which randomizes patients with an uneventful one year course after a DES implantation, to an additional year of clopidogrel and aspirin therapy versus aspirin alone, will be able to answer the important question about the role of extended (2y) dual anti-platelet therapy with clopidogrel and aspirin after DES implants. The investigators hypothesize that clopidogrel discontinuation at 1 year post-DES implantation is associated with an increase in cardiovascular events during the one year of follow-up period.

DETAILED DESCRIPTION:
SCORE is a multicenter, prospective randomized study of post-percutaneous coronary intervention (PCI) patients with an uneventful 1 year post-PCI course on dual anti-platelet therapy (DAPT) with clopidogrel and aspirin. Patient will be randomized to an additional 1 year of DAPT (treatment arm) vs. aspirin alone (control arm)to assess the following endpoints during the 1 year follow-up period:

1. Death / Myocardial infarction (MI) (Primary end-point)
2. Combined endpoints of death, myocardial infarction, repeat revascularization, stroke, and major/minor bleeding (Secondary end-point)

During the year of follow up, subjects will be contacted once every three months. This will enable us to track study endpoints in the study population. In addition the patients' medical records will be screened to investigate if any of the aforementioned endpoints have been reached.

ELIGIBILITY:
Inclusion Criteria:

* Post-PCI patients receiving at least 1 DES
* Completed 9-15 months follow-up free of MI, repeat revascularization
* Able to provide informed consent
* Have continued dual anti-platelet therapy with aspirin and clopidogrel for 1 year post-PCI

Exclusion Criteria:

* Patients allergic to aspirin
* Patients with aspirin resistance
* Patients with allergy to clopidogrel
* Patients on concomitant warfarin therapy
* History of bleeding diathesis, coagulopathy, and/or platelet count < 100,000 cubic mm
* Patients with a life expectancy less than 1 year due to active cancers (except basal cell carcinoma)
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-09-11 (Actual); Primary Completion 2014-03-03 (Actual); Study Completion 2014-03-03 (Actual)

PRIMARY OUTCOMES:
Death and Myocardial Infarction | 12 months

SECONDARY OUTCOMES:
Combined endpoints of death, myocardial infarction, repeat revascularization, stroke and major/minor bleeding | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — VA North Texas Healthcare System, UT Southwestern Medical Center; Emmanouil S Brilakis, MD, PhD, Study Director — VA North Texas Healthcare System, Dallas, TX
Locations (3):
- Dallas Veterans Hospital, Dallas, Texas, United States
- The Onassis cardiac Surgery Centre, Athens, Greece
- Escorts Health Institute & Research Centre Ltd, New Delhi, India

REFERENCES:
- [Background] Banerjee S, Varghese C, Samuel J, Weideman RA, Little BB, Kelly KC, Rao SV, Reilly RF, Brilakis ES. Comparison of the impact of short (<1 year) and long-term (> or =1 year) clopidogrel use following percutaneous coronary intervention on mortality. Am J Cardiol. 2008 Nov 1;102(9):1159-62. doi: 10.1016/j.amjcard.2008.06.058. Epub 2008 Sep 11. PMID 18940284
- [Background] Ho PM, Peterson ED, Wang L, Magid DJ, Fihn SD, Larsen GC, Jesse RA, Rumsfeld JS. Incidence of death and acute myocardial infarction associated with stopping clopidogrel after acute coronary syndrome. JAMA. 2008 Feb 6;299(5):532-9. doi: 10.1001/jama.299.5.532. PMID 18252883